CLINICAL TRIAL: NCT00001287
Title: The Efficacy of High-Dose Intravenous Immunoglobulin in Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: Intravenous Immunoglobulin (IVIg) for the Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 910039; 91-N-0039
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Demyelinating Diseases; Paraproteinemias
Keywords: Intravenous High-Dose Immunoglobulin; Monoclonal Gammopathies; Peripheral Nerve Demyelination; CIDP; Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Demyelinating Diseases; Paraproteinemias; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: intravenous immunoglobulin (IVIg)

SUMMARY:
Chronic Inflammatory Demylinating Polyneuropathy (CIDP) is an autoimmune condition affecting the nervous system. Researchers believe the immune system begins attacking the cells covering nerves called myelin. The destruction of myelin causes muscle weakness, loss of sensation, abnormal levels of protein in the fluid surrounding the brain (CSF), and slowing of the nervous system. The disease progresses slowly and disables patients suffering from it.

CIDP is treated with steroids, plasmapheresis, and immunosuppressive drugs. Many patients initially respond to these treatments, but develop resistance to the therapy or experience side effects causing the treatments to be stopped.

Researchers believe that intravenous immunoglobulin (IVIg) may provide patients with CIDP a safer and more effective alternative to standard therapies for the disease. IVIg is a drug that has been used successfully to treat other immune-related diseases of the nervous system. However, because IVIg is so expensive, researchers believe it should first be proven effective on a small group of patients.

The study will take 60 patients with CIDP and divide them into two groups. Group one will receive 2 injections of IVIg once a month for three months. Group two will receive 2 injections of placebo "inactive injection of sterile water" once a month for three months. Following the three months of treatment, group one will begin taking the placebo and group two will begin taking IVIg for an additional 3 months. The drug will be considered effective if patients receiving it experience a significant improvement (>25%) in muscle strength.

DETAILED DESCRIPTION:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a slowly progressive disabling neuropathy characterized by subacute onset of muscle weakness, distal sensory deficit, elevated spinal fluid protein, and slow nerve conduction velocity with or without conduction block. A monoclonal gammopathy is at times present in the serum of some patients. Because immune-mediated mechanisms against peripheral nerve myelin are thought to be primarily responsible for the clinical manifestations of CIDP, the treatment of choice is with corticosteroids, plasmapheresis or immunosuppressive drugs. Although many patients initially respond to these agents, a large number of them become resistant or develop unacceptable side effects that necessitate their discontinuation. The need for a more effective and safe immunotherapy in CIDP patients prompted the present study using high-dose intravenous immunoglobulin (IVIg). IVIg is an immunomodulating agent which has been recently shown to be effective and safe in the treatment of a number of patients with immune-related neuromuscular diseases.

This is a double blind, randomized, placebo controlled, trial involving 60 patients, half of which will receive IVIg and the other half placebo (D5/W). Because IVIg is prohibitively expensive, a controlled trial is needed to provide convincing evidence of efficacy, and ensure that the benefit is not due to spontaneous improvement or to observer bias. The dose of IVIg is 2 GM/Kg divided into two daily doses administered monthly for six months. The drug will be considered effective if patients experience an increase of more than 25% in their baseline muscle strength. Muscle strength will be assessed with a series of objective dynamometric measurements performed before and after each monthly infusion.

ELIGIBILITY:
Selected patients should have CIDP with or without an associated monoclonal gammopathy.

Subjects should have clinical evidence of peripheral neuropathy with muscle weakness and sensory deficit.

Subjects should have evidence of clinical, histological or family history of another neuromuscular illness.

Subjects should have elevation of CSF protein during the course of the disease.

Subjects should have demyelination by nerve conduction study and/or nerve biopsy.

Suitable candidates for IVIg should be patients with active, bonefide CIDP who:

1. have been treated with steroids but had: a) no response or incomplete response (as defined by continued muscle weakness) to high-dose therapy or b) a good response to steroids but inability to taper the dose without a flare of disease activity or c) unacceptable steroid side effects such as gastrointestinal hemorrhages, osteonecrosis, hyperglycemia, extreme weight gain etc. or
2. have been additionally treated with one of the other immunosuppressive agents considered effective in some CIDP patients, such as azathioprine, chlorambucil, cyclophosphamide, cyclosporine or plasmapheresis but without benefit or with unacceptable side effects that had necessitated their discontinuation.

Subjects should not be pregnant or nursing.

Subjects should not be critically ill such as those requiring intravenous pressors for maintenance of cardiac output, patients with unstable respiratory insufficiency and patients with such severe muscle weakness requiring help for basic self care (Karnofsky performance scale less than 50).

No subjects below 18 years of age.

Patients should not have severe renal or hepatic disease and severe COPD or coronary artery disease.

Patients should not be allergic to IVIg or have a known IgA deficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1990-12; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dalakas MC, Engel WK. Chronic relapsing (dysimmune) polyneuropathy: pathogenesis and treatment. Ann Neurol. 1981;9 Suppl:134-45. doi: 10.1002/ana.410090719. PMID 7224612
- [Background] Cook D, Dalakas M, Galdi A, Biondi D, Porter H. High-dose intravenous immunoglobulin in the treatment of demyelinating neuropathy associated with monoclonal gammopathy. Neurology. 1990 Feb;40(2):212-4. doi: 10.1212/wnl.40.2.212. PMID 2153942
- [Background] Basta M, Dalakas MC. High-dose intravenous immunoglobulin exerts its beneficial effect in patients with dermatomyositis by blocking endomysial deposition of activated complement fragments. J Clin Invest. 1994 Nov;94(5):1729-35. doi: 10.1172/JCI117520. PMID 7962520